CLINICAL TRIAL: NCT05546294
Title: The Effects of Aerobic Exercise on Sleep Quality, Fatigue, Quality of Life, Depression, Serum BDNF and Irisin Levels in Patients With Rheumatoid Arthritis: A Prospective Randomized Controlled Study
Brief Title: The Effects of Exercise on Serum BDNF and Irisin Levels in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Hatice Kudret Miroğlu, Research Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAİRİSİNBDNF2021
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis; Sleep Quality; Aerobic Exercise
Keywords: Rheumatoid Arthritis; Sleep Quality; Serum BDNF; Serum Irisin; Quality of Life; Fatigue; Depression
MeSH Terms: conditions — Arthritis, Rheumatoid; Sleep Initiation and Maintenance Disorders; Fatigue; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RA patients receiving aerobic and home exercise (Experimental): A total of 20 sessions of aerobic exercises using bicycle ergometer, five times a week and once a day for four weeks, were applied to the patients. Then the patients were showed a daily home exercise program to apply once a day at their home.
  Interventions: Device: Aerobic and home exercise
- RA patients receiving only home exercise (Active Comparator): The patients were showed only a daily home exercise program to apply once a day at their home.
  Interventions: Other: Home exercise
- Healthy control group (Other): There is no intervention to this group.
  Interventions: Other: Healthy control group

INTERVENTIONS:
Device: Aerobic and home exercise — A total of 20 sessions of aerobic exercises using bicycle ergometer, five times a week and once a day for four weeks, were applied to the patients.Maximum heart rate was calculated for each subject (220 - age) and a heart rate monitor will be used to follow subjects' heart rate during aerobic exercise.
  Then the patients were showed a daily home exercise program to apply once a day at their home.
  As a daily home exercise program:ROM exercises and strengthening exercises for major muscle groups (such as abdominal muscles, erector spinae, hamstring, quadriceps, hip flexors, strengthening exercises for all extremities) were showed.
  At the beginning of the treatment and at the end of the treatment (4th week), serum BDNF and irisin levels will be tested using the ELISA kit, with blood samples taken from the RA patients in the early morning.
  Arms: RA patients receiving aerobic and home exercise
Other: Home exercise — The patients were showed only a daily home exercise program to apply once a day at their home.
  As a daily home exercise program:ROM exercises and strengthening exercises for major muscle groups (such as abdominal muscles, erector spinae, hamstring, quadriceps, hip flexors, strengthening exercises for all extremities) were showed.
  At the beginning of the treatment and at the end of the treatment (4th week), serum BDNF and irisin levels will be tested using the ELISA kit, with blood samples taken from the RA patients in the early morning.
  Arms: RA patients receiving only home exercise
Other: Healthy control group — Serum BDNF and irisin levels will be tested using the ELISA kit, with blood samples taken only once from healthy control group in the early morning. It will be checked whether there is a difference between the basal serum BDNF and irisin levels of rheumatoid arthritis patients and healthy control group.
  Arms: Healthy control group

SUMMARY:
The aim of our study is to investigate the effects of aerobic exercise on sleep quality, fatigue, quality of life, depression and serum BDNF and irisin levels, which are important biomarkers of sleep in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, progressive, autoimmune disease characterized primarily by inflammation of synovial joints and tendon sheaths of synovial nature.

Sleep disturbance in RA patients has a negative impact on their quality of life in addition to their mental and physical health. Exercise has been identified as an important non-pharmacological factor in improving sleep quality and mood in patients with rheumatoid arthritis.

Irisin is a myokine and adipokine that has anti-inflammatory effects and can help regulate energy expenditure. It is secreted from skeletal muscles after exercise, as well as from other tissues such as the liver, nerves, heart, kidneys and skin. It has been observed that serum irisin levels are decreased in RA patients with poor sleep quality compared to RA patients with good sleep quality.

BDNF, one of the biochemical parameters evaluating sleep, is a signal protein encoded by the BDNF gene located on chromosome 11. It belongs to the neurotrophin family, which regulates the survival, development and function of neurons. Neuronal activity is a powerful stimulant that elicits BDNF production. Thus, activation of brain areas associated with motor control during exercise contributes to increased BDNF production in the brain and additionally in plasma. During acute exercise, irisin stimulates BDNF expression in the hippocampus of the brain. In addition to the circadian variation of plasma BDNF, the blood concentration of BDNF has been shown to increase acutely in response to aerobic exercise that does not include resistance exercise. Moreover, it has been reported that people with higher basal serum BDNF concentrations have lower REM sleep and therefore less sleep disturbances.

This investigation was designed as prospective randomized controlled study. Participants were randomized into 3 groups; RA patients receiving aerobic and home exercise, RA patients receiving only home exercise and healthy control group.

As evaluation parameters, DAS28 Score, SF (Short form) -36 Quality of Life Scale, Pittsburgh Sleep Quality Index (PSQI), Fatigue Severity Scale (FSS), Beck Depression Inventory (BDI), 6 Minute Walk Test and Borg Scale will be evaluated with. It was planned that the evaluations were made and recorded by a blinded physician to the all patients with rheumatoid arthritis at the beginning of the treatment and at the end of the treatment.In the healthy control group, the evaluation parameters will be examined only once at the beginning of the study.

At the beginning of the treatment and at the end of the treatment (4th week), serum BDNF and irisin levels will be tested using the ELISA kit, with blood samples taken from the RA patients in the early morning. It will be checked whether there is a difference between the basal serum BDNF and irisin levels of rheumatoid arthritis patients with the blood sample taken only once in the early morning from the healthy control group.

ELIGIBILITY:
Inclusion Criteria: Patients were included in the study

* Male and female gender between the ages of 20 and 60 who were diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR diagnostic criteria,
* Patients with Disease Activity Score (DAS28) ≤3.2 (low disease activity or remission) (no change in anti-rheumatic drugs or steroid dose in the last 3 months),
* Patients who were being followed at Afyonkarahisar Health Sciences University Department of Physical Medicine and Rehabilitation,

Exclusion Criteria:

* Active malignancy and/or a history of malignancy within the past 5 years,
* Uncontrolled cardiopulmonary disease (such as severe hypertension, chronic obstructive pulmonary disease, stage 3 or 4 heart failure, significant left ventricular outflow obstruction, dissecting aneurysm, embolism or thrombophlebitis history),
* Patients who cannot tolerate cardiorespiratory exercise training due to unstable angina pectoris, dangerous cardiac arrhythmias and myocardial infarction in the last 3 months,
* Pregnancy or planning a pregnancy in the near future,
* History of major surgery (including joint surgery) within the last six months,
* Regular physical activity at least 3 days a week in the last 3 months,
* Orthopedic, neurological or mental disease that may affect exercise,

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline disease activity score (DAS28) at 4th week | Up to 4th week
  DAS 28 is a scale consisting of 4 parameters; tender and swollen joint counts from 28 joints (shoulders, elbows, wrists, MCFs,PIPs and knee joints), blood sedimentation (mm/hour) or CRP (mg/liter) value and patient global assessment (between 0 and 100; Best imaginable health condition-100, The worst possible health condition -0) A mathematical formula is used to calculate the overall score. DAS28 can range from 0 to 9.4.Generally, a DAS28 score of;
  * More than 5.1 indicates high disease activity
  * Between 3.2 and 5.1 indicates moderate disease activity
  * Between 2.6 and less than 3.2 indicates low disease activity
  * Lower than 2.6 indicates disease remission
  It is only applied to Rheumatoid Arthritis patients.

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36 (SF-36)) at 4th week | Up to 4th week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
  It is applied to all RA patients at the baseline and 4th week, and only applied once to healthy control group at the baseline.
Change from baseline Fatigue Severity Scale (FSS) at 4th week | Up to 4th week
  The scale evaluates the fatigue severity of the participants in the last week. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. The minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities.
  It is applied to all RA patients at the baseline and 4th week, and only applied once to healthy control group at the baseline.
Change from baseline Beck's Depression Inventory (BDI) at 4th week | Up to 4th week
  The Beck Depression Inventory (BDI) is a 21-item (Each question had a set of at least four possible responses, ranging in intensity), self-report rating inventory that measures characteristic attitudes and symptoms of depression. It is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex.
  * 0-9: indicates minimal depression
  * 10-18: indicates mild depression
  * 19-29: indicates moderate depression
  * 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
  It is applied to all RA patients at the baseline and 4th week, and only applied once to healthy control group at the baseline.
Change from baseline Pittsburgh Sleep Quality Index (PSQI) at 4th week | Up to 4th week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval.Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
  It is applied to all RA patients at the baseline and 4th week, and only applied once to healthy control group at the baseline.
Change from baseline Six Minute Walk Test (6MWT) at 4th week | Up to 4th week
  Walking distance, starting and ending blood pressure, heart rate, and oxygen saturation values will be recorded by applying a 6-minute walking test in a 40-meter corridor to the patients who will be applied bicycle ergometry.
  It is only applied to RA patients receiving aerobic exercise.
Change from baseline Borg Rating Of Perceived Exertion Scale (Borg RPE Scale) at 4th week | Up to 4th week
  Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. It is a scale of 6-20; it has a high correlation to heart rate and multiplying each number by 10 gives the training heart rate as at the time of scoring.
  In Borg RPE;
  * 9 = 'very light' exercise which equals walking slowly for a few minutes at the own pace of a healthy individual.
  * 13 = 'somewhat hard' but the individual is still able to continue the activity.
  * 17 = 'very hard'. A healthy person can continue but must push themselves beyond their comfort of being very fatigued.
  * 19 = extremely strenuous exercise.for most people, the hardest they have ever experienced.
  It is only applied to RA patients receiving aerobic exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Ümit DÜNDAR, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Hatice Kudret MİROĞLU, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baillet A, Zeboulon N, Gossec L, Combescure C, Bodin LA, Juvin R, Dougados M, Gaudin P. Efficacy of cardiorespiratory aerobic exercise in rheumatoid arthritis: meta-analysis of randomized controlled trials. Arthritis Care Res (Hoboken). 2010 Jul;62(7):984-92. doi: 10.1002/acr.20146. PMID 20589690
- [Background] Gamal RM, Mohamed ME, Hammam N, El Fetoh NA, Rashed AM, Furst DE. Preliminary study of the association of serum irisin levels with poor sleep quality in rheumatoid arthritis patients. Sleep Med. 2020 Mar;67:71-76. doi: 10.1016/j.sleep.2019.10.021. Epub 2019 Nov 30. PMID 31918120
- [Background] Tan X, van Egmond LT, Cedernaes J, Benedict C. The role of exercise-induced peripheral factors in sleep regulation. Mol Metab. 2020 Dec;42:101096. doi: 10.1016/j.molmet.2020.101096. Epub 2020 Oct 9. PMID 33045432